CLINICAL TRIAL: NCT06583642
Title: Antimicrobial Therapeutic Drug Monitoring During Lung Transplant Perioperative Phase
Status: Not yet recruiting | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Giacomo Grasselli, MD, Policlinico Hospital
Other Study IDs: ATB_LuTx
Record Dates: First submitted 2024-09-01; First posted 2024-09-04 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Lung Transplant Infection; Pneumonia, Bacterial; Antibiotic Resistant Strain
MeSH Terms: conditions — Pneumonia, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected: at ICU admission, the first morning after LuTx and at 72h after LUTX. Each blood sample (4 mL) will be centrifuged, and plasma samples stored at -20°C until analysis;
  Bronchoalveolar lavage samples will be collected exclusively first morning after LuTx and at 72h after LUTX. Each BAL sample (4 mL) will be centrifuged, and supernatant samples stored at -20°C until analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background: Post-LUTX pneumonia represents a leading cause of death along the first month after LUTX. Donor-derived transmission of pathogenic species occurs up to 25% of recipients receiving a graft with a positive BAL culture, despite in-vitro adequate antimicrobial prophylaxis.

Hypothesis: LUTX recipients are either exposed to suboptimal antimicrobial doses or antimicrobial penetration into the lug parenchyma is altered either due to surgery (absence of bronchial anastomoses) or to the hyperinflammatory state.

Methods: LUTX recipients admitted to the intensive care unit at the Fondazione IRCCS Ca' Granda Policlinico Hospital. According to the institutional perioperative prophylaxis protocol and the donor/recipient ecology the most frequent antimicrobial molecules administered will be: cefepime, vancomycin, and meropenem. Antimicrobial pharmacokinetics will be investigated at three timepoints. Plasma levels of the ongoing antimicrobial molecule will be assessed at ICU admission, on postoperative day 1 and on postoperative day 3. Bronchoalveolar lavage (BAL) samples for the measurement of BAL antimicrobial levels will be collected during the BAL performed for clinical indication on postoperative day 1 and on postoperative day 3.

Absolute plasma and BAL antimicrobial levels will be assessed. The ratio of BAL to plasma dosage of antimicrobial will be assessed to evaluate antimicrobial penetration within the target tissue. Correlation between both plasma and BAL antimicrobial dosage and recipients' postoperative fluid balance, body weight, vasopressor requirement, renal function will be performed.

DETAILED DESCRIPTION:
1. BACKGROUND

   Lung Transplantation (LUTX) is the curative treatment for selected patients with end-stage lung disease. Despite continuous optimization of recipients perioperative phase morbidity and mortality remain about 20%. Bacterial infections are a leading cause of death in the early post-transplant period.

   Donor-recipient transmission of pathogens plays an actual role in worsening graft function. The rate of donor with bacterial growth on the pre-LUTX bronchoalveolar lavage (BAL) is high (36%).Furthermore, among uncolonized recipients, receiving a graft with a positive BAL carries the risk of developing a donor-derived infection (DDI) in almost one quarter of cases, affecting early graft function, despite recipients were already treated with an "in-vitro appropriate" antibiotic therapy. In this scenario, the adequacy of perioperative antimicrobial prophylaxis might play a major in preventing either donor derived pulmonary or surgical site infections.

   Aim of the present study is to describe the PK of the most frequently used perioperative antimicrobials (i.e., cefepime, meropenem, and vancomycin) in plasma and in the bronchoalveolar lavage of patients undergoing double LUTX during the immediate postoperative phase.
2. HYPOTHESIS of the study

Hypothesis of the study is that LUTX recipients are either exposed to suboptimal antimicrobial doses or antimicrobial penetration into the lug parenchyma is altered either due to surgery (absence of bronchial anastomoses) or to the hyperinflammatory state.

Objective of the study is to describe and model the PK of cefepime, meropenem, and vancomycin in adult patients undergone primary double LUTX.

3 METHODS

Prospective observational single-center pharmacological biological no-profit study.

3.1 Primary Endpoints PK/PD of cefepime, vancomycin and meropenem in adult patients undergone primary double lung transplant.

3.2 Secondary Endpoints

1. To measure the ratio between BAL fluid and plasma antibiotic level of antimicrobials in order to quantify the antimicrobial penetration into the lung tissue
2. To identify the clinical factors correlated to subtherapeutic suboptimal exposure of antimicrobials in LUTX recipients perioperative phase

3.3 Setting The study will be carried out in the Institutional ICU (General Intensive Care Unit, E.Vecla), as well as the thoracic surgery and pneumology unit.

4 PROCEDURES

Participation in the study will not change the standard enlistment protocol, the surgery procedure, or anesthesiologic management.

4.1 Drug Administration

All the patients will be treated as per standard clinical management. In particular, vancomycin, cefepime, and meropenem will be provided to the patients as per their international approved and Italian (Agenzia Italiana del Farmaco) indications, following their drug information leaflet, at discretion of the caring physician.

In particular:

* Cefepime represents the Institutional molecule of choice for perioperative prophylaxis. A loading dose of 2g is administered before surgical incision and repeated every 4 hours along surgery. Additional 1g dose is administered whenever severe bleeding (>1.5Lt) occurs or ECMO support is required. Postoperatively, at ICU admission, a continuous infusion of 6g/day is started and then prosecuted, stopped or modified according to the result of the mPCR on BAL performed on the 3rd postoperative day. Dose adjustment will be performed by the treating physician according to daily measured patients' creatinine clearance.
* Vancomycin is administered before surgical incision at a dose 15mg/Kg and not repeated throughout surgery. Whenever either donor or recipient BAL will test positive for methicillin resistant staphylococcus aureus Vancomycin treatment will be started at a dose of 25mg/kg loading dose followed by continuous infusion of 20mg/kg. Daily plasma level will be assessed by the treating physician and dose adjustment will be performed accordingly.
* Meropenem will be started whenever either the donor or the recipient's BAL will test positive for CTX-M mechanism of antimicrobial resistance. Meropenem will be administered with a loading dose of 2g followed by a continuous infusion of 6g/day. Dose adjustment will be performed by the treating physician according to daily measured patients' creatinine clearance.

4.2 Study Procedures

Once admitted to the Intensive Care Unit patients a continuous infusion of cefepime (6g/day) will be started. A 4 ml blood sample remnant (from the daily blood lab tests performed in the ICU) will be collected for the measurement of antimicrobial plasma level immediately after surgery. The blood sample will be centrifuged at 4°C, 3000 rpm for 15 min. Plasma sample, collected in a deidentified cryovial, will be stored at -80°C in a refrigerator located in the Intensive Care Unit. Simultaneously, measurement of patient weight, arterial and venous blood gas analysis (to calculate intrapulmonary shunt) and lung mechanics (i.e. static lung compliance) will be performed.

Similarly the first morning and at 72h after LUTX, the thoracic surgeon will perform a bronchoscopy to check for the integrity of bronchial anastomosis and will perform a surveillance BAL which will be processed for both fast and standard microbiological tests. At each BAL performed 4 mL of discard BAL sample will be collected for the measurement of BAL antimicrobial level. Simultaneously to the BAL, a 4 ml blood sample remnant (from the daily blood lab tests performed in the ICU) will be collected for the measurement of antimicrobial plasma level. The blood sample will be centrifuged at 4°C, 3000 rpm for 15 min. Plasma sample, collected in a deidentified cryovial, will be stored at -80°C in a refrigerator located in the Intensive Care Unit. Simultaneously, measurement of patient weight, arterial and venous blood gas analysis (to calculate intrapulmonary shunt) and lung mechanics (i.e. static lung compliance) will be performed. Renal function (i.e. creatinine clearance and fraction of excreted urea and sodium), measured daily in the Intensive Care Unit, will be collected. A chest X-Ray, performed per clinical practice to grade Primary graft dysfunction at 24 and 72 hours after LUTX, will be collected.

In summary, to carry out the PK study, we will collect a total amount of 12 mL of blood, and 8 mL of bronchoalveolar lavage. Those samples will be transferred to the collaborating center (Ospedale Luigi Sacco), and analyzed for PK study, as follows:

* Blood samples will be collected: at ICU admission, the first morning after LuTx and at 72h after LUTX. Each blood sample (4 mL) will be centrifuged, and plasma samples stored at -20°C until analysis;
* Bronchoalveolar lavage samples will be collected exclusively first morning after LuTx and at 72h after LUTX. Each BAL sample (4 mL) will be centrifuged, and supernatant samples stored at -20°C until analysis.

Thus, cryopreserved samples will be shipped to the collaborating center (ASST Fatebenefratelli Sacco, University Hospital, Milan, Italy) at the end of the recruitment period, and thus tests will be performed. The antibiotic concentrations will be determined using an ultra-performance liquid chromatography-tandem mass spectrometry method (LC-MS/MS). After purification through precipitation and dilution with a solution of methanol, acetonitrile, and water with 0.1% formic acid, 1µL will be injected. The chromatographic separation will be achieved using a gradient (acetonitrile and water with formic acid 0.1%) on a reversed-phase analytical column (acuity UPLC BEH C18 1.70lm2.1%50mm; Waters, Milan, Italy). For quantification, the analysis will be performed in ESI-positive mode. Then, PK modeling will be carried out as previously done by the collaborating center.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of LUTX
* Age > 18 years
* Signed informed consent

Exclusion Criteria:

* Age < 18 years old
* Already undergone LUTX
* Documented respiratory colonization in the 12 months preceding LUTX
* Undergoing any antimicrobial therapy preceding LUTX
* Documented post-LUTX endobronchial plasma leak requiring high levels of PEEP > 15 cmH2O.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise adult patients undergone primary double lung transplant without pre-operative lung colonization, and undergoing perioperative antibiotic therapy with cefepime, or meropenem.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Plasma Antimicrobial Concentration | ICU admission after LuTX; 12 hours after LuTX; 72 hours after LuTX
  Dosage of plasma levels of Cefepime or Meropenem or Vancomycin
Bronchoalveolar Antimicrobial Concentration | ICU admission after LuTX; 12 hours after LuTX; 72 hours after LuTX
  Dosage of bronchoalveolar levels of Cefepime or Meropenem or Vancomycin
Antimicrobial lung tissue penetration | ICU admission after LuTX; 12 hours after LuTX; 72 hours after LuTX
  Ratio of bronchoalveolar to plasma concentration of Cefepime or Meropenem or Vancomycin

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca'Granda - Ospedale Maggiore Policlinico, Milan, Milan, Italy